CLINICAL TRIAL: NCT02657915
Title: A Multicenter, Follow-Up Study to Assess Long-Term Electrophysiologic and Clinical Outcomes in Subjects Previously Enrolled in Study 215ON201
Brief Title: Long-Term Assessment of Remyelinating Therapy
Acronym: RENEWED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 215ON203; 2015-003618-26 (EudraCT Number)
Record Dates: First submitted 2015-12-23; First posted 2016-01-18 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Acute Optic Neuritis
Keywords: FF-VEP; mfVEP; Human anti-LINGO-1; BIIB033; AON
MeSH Terms: interventions — Sodium Chloride; Organization and Administration; opicinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This was a follow-up study with no investigational product; however, the allocation method in RENEW Study (NCT01721161) was randomised-controlled and to maintain the blind from RENEW, the treatment disclosure for RENEW was not shared with study sites or participants until the end of this study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): This was a follow-up study, investigational product was administered in the previous study. Participants in the placebo arm have received at least 1 dose of placebo.
  Interventions: Drug: Placebo
- BIIB033 100mg/Kg (Experimental): This was a follow-up study, investigational product was administered in the previous study. Participants in the BIIB033 arm have received at least 1 dose of 100 mg/kg BIIB033.
  Interventions: Drug: BIIB033 100mg/Kg

INTERVENTIONS:
Drug: Placebo — Administered as specified in the treatment arm.
  Other Names: Sterile normal saline (0.9% sodium chloride for IV administration)
  Arms: Placebo
Drug: BIIB033 100mg/Kg — Administered as specified in the treatment arm.
  Arms: BIIB033 100mg/Kg

SUMMARY:
The primary objective of the study is to assess full-field visual evoked potential (FF-VEP) latency in subjects who were enrolled in Study NCT01721161 2 years (+ up to 12 months) after the last study visit. The secondary objective is to assess clinical progression and severity of central nervous system (CNS) demyelinating disease in subjects who were enrolled in Study NCT01721161 2 years (+ up to 12 months) after the last study visit. Intervention was administered in the previous study. The participants, investigator and outcome assessors remain blinded in this follow-up study.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have participated in Study NCT01721161 and received at least 1 dose of BIIB033 or placebo, as per protocol, within 2 years (+ 4 months) from Day 1 of this study (2 years from Week 32 or projected Week 32 visit, if the subject did not complete all visits in Study NCT01721161).

Key Exclusion Criteria:

* Not previously enrolled in Study NCT01721161
* Subjects with recent kidney function, such as serum creatinine above upper limit of normal range, will not be allowed to receive administration of Gd but will otherwise be allowed to participate in the study, including magnetic resonance imaging (MRI) assessments not requiring the use of Gd.
* Female subjects must have had a recent pregnancy test and must not be breastfeeding prior to MRI assessments with Gd.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (23):
- Australia (2):
  - Research Site, Sydney, New South Wales
  - Research Site, Parkville, Victoria
- Research Site, Bruges, Belgium
- Research Site, Ottawa, Ontario, Canada
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Glostrup Municipality, Denmark
- Germany (5):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Tübingen
- Research Site, Budapest, Hungary
- Research Site, Milan, Italy
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Murcia
  - Research Site, Seville
  - Research Site, Valencia
- Research Site, Solna, Sweden
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants eligible for this study was determined by the number of participants who participated in RENEW Study (NCT01721161). A total of 82 participants were enrolled in RENEW Study (NCT01721161) and received at least 1 dose of study treatment. A total of 52 participants participated in this study.
Groups:
- Placebo: This was a follow-up study with no investigational product administered. Participants in the placebo arm had received at least 1 dose of placebo in RENEW Study (NCT01721161).
- BIIB033 (Opicinumab) 100 mg/kg: This was a follow-up study with no investigational product administered. Participants in the BIIB033 (Opicinumab) arm had received at least 1 dose of 100 milligram per kilogram (mg/kg) BIIB033 in RENEW Study (NCT01721161).
Period: Overall Study
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Started | 24 | 28
Intent-to Treat (ITT) Population | 24 | 28
Per-protocol Population | 23 | 24
Completed | 24 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all randomized participants who received at least 1 dose of study treatment in RENEW Study (NCT01721161) and completed at least 1 of the Day 1 assessments in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (7.96) | 34.6 (6.57) | 35.1 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Reason for Not Reporting category of Race/Ethnicity is confidentiality regulations.
  Participants
    White | 4 | 4 | 8
    Not reported | 20 | 24 | 44

OUTCOME MEASURES:

1. Primary Outcome: FF-VEP Latency of the Affected Eye as Compared to the Baseline of the Fellow Eye at 2 Years (+ up to 12 Months) After the Last Study Visit Assessment (Week 32) in RENEW Study (NCT01721161)
Description: A full field visual evoked potential (FF-VEP) is an evoked potential caused by a visual stimulus, such as an alternating checkerboard pattern on a computer screen. Responses are recorded from electrodes that are placed on the back of the head and are observed as a reading on an electroencephalogram (EEG). These responses usually originate from the occipital cortex, the area of the brain involved in receiving and interpreting visual signals.
Time Frame: Baseline (RENEW Study [NCT01721161]), Day 1 (NCT02657915)
Population: Per protocol (PP) population: defined as participants from ITT population who completed the study, did not miss more than 1 dose of BIIB033 (Opicinumab) or placebo, and did not receive MS modifying therapies in RENEW Study (NCT01721161). The statistical analysis plan specified that efficacy analyses performed in PP were considered primary analyses.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
milliseconds (msec)
  Baseline: number analyzed (Participants) | 22 | 24
  Baseline | 100.68 (4.854) | 102.29 (5.507)
  Day 1: number analyzed (Participants) | 21 | 23
  Day 1 | 119.52 (13.395) | 114.20 (14.235)
Statistical Analysis 1: Comparison: Placebo vs BIIB033 (Opicinumab) 100 mg/kg; Test type: Superiority; p = 0.165, ANCOVA; Mean Difference (Final Values) = -6, 95% CI 2-sided [-14.56 to 2.57]

2. Secondary Outcome: Number of Participants That Developed Clinically Definite Multiple Sclerosis (CDMS) After Enrollment in RENEW Study (NCT01721161)
Description: The diagnosis of clinically definite multiple sclerosis (CDMS) was made on the basis of clinical criteria and requires that a patient experience at least 2 neurologic events consistent with demyelination, separated both in time and in location in the central nervous system.
Time Frame: RENEW Study (NCT01721161) to Day 1 (NCT02657915)
Population: The PP population was defined as participants from the ITT population who completed the study, did not miss more than one dose of BIIB033 (Opicinumab) or placebo, and did not receive MS modifying therapies in RENEW Study (NCT01721161).
Measure: Number; unit: participants
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
participants | 12 | 12

3. Secondary Outcome: Time to Diagnosis of CDMS
Description: The diagnosis of CDMS was made on the basis of clinical criteria and requires that a patient experience at least 2 neurologic events consistent with demyelination, separated both in time and in location in the central nervous system. Time to diagnosis of CDMS in Study NCT02657915 was the time from the diagnosis of acute optic neuritis (AON) to the date of confirmed MS. Measured in Days using the Median (50th percentile) for each arm.
Time Frame: RENEW Study (NCT01721161) to Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
days | 386.0 [212.0 to 1065.0] | 909.5 [281.0 to NA] — Data was not reported for this value as it was not observed during this study.

4. Secondary Outcome: Severity of Central Nervous System (CNS) Demyelinating Disease as Assessed Using the Expanded Disability Status Scale (EDSS)
Description: The EDSS score is based on neurological testing and an examination of functional systems (FS), which are areas of the central nervous system which control bodily functions. These functional systems are: pyramidal (ability to walk), Cerebellar (coordination), brain stem (speech and swallowing), sensory (touch and pain), bowel and bladder functions, visual, mental and Other (includes any other neurological findings due to MS). An overall score ranging from 0 (normal) to 10 (disability) was calculated. Higher scores indicate greater disability.
Time Frame: Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
score on a scale | 1.22 (0.837) | 1.26 (1.136)

5. Secondary Outcome: Severity of CNS Demyelinating Disease as Assessed Using the Symbol- Digit Modalities Test (SDMT)
Description: SDMT is a screening test for cognitive impairment. Participants were given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best). Originate from the occipital cortex, the area of the brain involved in receiving and interpreting visual signals.
Time Frame: Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
score on a scale | 56.7 (9.91) | 58.7 (9.01)

6. Secondary Outcome: Severity of CNS Demyelinating Disease as Assessed Using the Multiple Sclerosis Functional Composite (MSFC) Assessment
Description: MSFC has 3 component- timed 25-foot walk (T25FW), 9-hole peg test (9HPT) [dominant and nondominant hands] and (3-second) paced auditory serial addition Test (PASAT). The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. MSFC Z-score = (Z25-foot-walk + Z9HPT + ZPASAT-3)/3, where Zj refers to Z-scores of component j. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Time Frame: Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
Z-score | -0.82 (2.883) | -0.06 (0.804)

7. Secondary Outcome: Change in Number of Gadolinium (Gd)-Enhanced Lesions From Baseline in RENEW Study (NCT01721161) to Day 1 (NCT02657915)
Description: Change in disease activity from baseline with brain magnetic resonance imaging (MRI) was calculated and reported. MRI analysis included number of consensus GD-enhanced lesions as a measure of disease activity.
Time Frame: Baseline (RENEW Study [NCT01721161]), Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
lesions
  Baseline: number analyzed (Participants) | 22 | 24
  Baseline | 0.2 (0.69) | 0.1 (0.41)
  Change at Day 1: number analyzed (Participants) | 21 | 19
  Change at Day 1 | 0.2 (1.54) | -0.1 (0.46)

8. Secondary Outcome: Change in Volume of T2 Lesions From Baseline in RENEW Study (NCT01721161) to Day 1 (NCT02657915)
Description: Change in disease activity from baseline with brain magnetic MRI was calculated and reported. MRI analysis included volume of T2 lesions as disease activity.
Time Frame: Baseline (RENEW Study [NCT01721161]), Day 1 (NCT02657915)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millilitres (mL)
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
Number analyzed (Participants) | 23 | 24
millilitres (mL)
  Baseline: number analyzed (Participants) | 22 | 24
  Baseline | 0.9710 (0.93551) | 0.7341 (1.29222)
  Change at Day 1: number analyzed (Participants) | 21 | 19
  Change at Day 1 | 0.5090 (1.38861) | 0.6244 (0.74850)

ADVERSE EVENTS:
Time Frame: Day 1 (NCT02657915)
Description: The safety population was defined as all participants who received at least 1 dose of study treatment in RENEW Study (NCT01721161) and completed at least 1 of the 1-day assessments in this study.
Arm/Group | Placebo | BIIB033 (Opicinumab) 100 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT02657915/SAP_000.pdf
  • Study Protocol (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02657915/Prot_001.pdf